CLINICAL TRIAL: NCT02209402
Title: Effect of a 3-month Aerobic Training Program on Endothelial Function in Mild-to-moderate CKD: a Randomized Controlled Trial
Brief Title: ENdothelial DysfUnction in Renal Disease and Exercise Training
Acronym: Endure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Amaryllis Van Craenenbroeck, Dr., Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EC/11/37/257
Record Dates: First submitted 2014-07-26; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Usual Care (No Intervention)
- Exercise Training (Experimental)
  Interventions: Behavioral: Exercise Training

INTERVENTIONS:
Behavioral: Exercise Training — Home-based training programme consisting of daily 4x10 minutes physical exercise on a magnetically braked bicycle at a heart rate corresponding to 80-90% of the heart rate achieved at the anaerobic threshold.
  Arms: Exercise Training

SUMMARY:
Chronic kidney disease (CKD) is a prevalent disorder and a major health concern. Cardiovascular disease is the most prevailing and life-threatening complication observed in patients with CKD. The diagnosis of CKD places a patient at the highest cardiovascular risk level irrespective of the stage of renal decline. Therefore, fatal cardiovascular events are more likely to occur than the evolution to final stages of kidney disease with the need for dialysis. Counter intuitively, treatment of classical cardiovascular risk factors does not affect cardiovascular prognosis in CKD, which suggests that the missing link between these two entities has not been elucidated yet.

In the present project, the investigators focus on endothelial dysfunction in patients with CKD. Endothelial dysfunction precedes overt atherosclerotic changes by many years. In the absence of structural changes, endothelial dysfunction is still reversible, which offers therapeutic perspectives to tackle the progression towards atherosclerosis in an early stage.

The purpose of this study is to determine whether an exercise training program is effective in ameliorating endothelial dysfunction in patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* patients with CKD stage 3-4 (eGFR (15-59 ml/min/1.73m2) without cardiovascular disease.

Exclusion Criteria:

* patients < 18 years
* pregnancy
* warfarin therapy
* glucocorticoid therapy
* clinically active malignant disease
* heart failure (ejection fraction < 50%)
* peripheral vascular disease, defined as a history of intermittent claudication, abnormal peripheral angiography or Doppler ultrasound, lower limb artery bypass surgery/angioplasty/stenting or non-traumatic lower extremity amputation
* cerebrovascular disease, defined as a history of transient ischemic attack (TIA) or stroke, significant stenosis of the A. carotis on ultrasound/CT angiography or carotid endarterectomy/stenting
* coronary artery disease (CAD), defined as a history of myocardial infarction, coronary artery angioplasty/stenting/bypass surgery, significant structural coronary lesions on angiography or high suspicion of CAD on a maximal exercise test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in brachial artery flow-mediated dilation (FMD= percentage constriction from baseline diameter to minimal occlusion diameter) | 3 months

SECONDARY OUTCOMES:
change in peak oxygen consumption (ml/kg/min) as marker of aerobic capacity | 3 months
change in aortic-femoral pulse wave velocity (m/s) as a marker of arterial stiffness | 3 months
change in augmentation index (%) as a marker of arterial stiffness | 3 months
change in Intima Media Thickness (µm) of the right common carotid artery | 3 months

OTHER OUTCOMES:
change in circulating endothelial progenitor cells (cells/1 million CD45+ events) | 3 months
change in migratory function of circulating angiogenic cells | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Antwerp, Antwerp, Belgium

REFERENCES:
- [Derived] Van Craenenbroeck AH, Van Craenenbroeck EM, Van Ackeren K, Vrints CJ, Conraads VM, Verpooten GA, Kouidi E, Couttenye MM. Effect of Moderate Aerobic Exercise Training on Endothelial Function and Arterial Stiffness in CKD Stages 3-4: A Randomized Controlled Trial. Am J Kidney Dis. 2015 Aug;66(2):285-96. doi: 10.1053/j.ajkd.2015.03.015. Epub 2015 May 8. PMID 25960303